CLINICAL TRIAL: NCT05106595
Title: Use of a Bimanual Arm Training Device in Acute Inpatient Stroke Rehabilitation, a Pre-post Cohort Study
Brief Title: Bimanual Arm Training in Acute Stroke
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00303045
Record Dates: First submitted 2021-10-20; First posted 2021-11-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Stroke, Acute; Upper Extremity Paresis
Keywords: rehabilitation; Occupational Therapists; Physical Therapists
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Traditional Occupational Therapy: participants receiving traditional occupational therapy treatments and interventions provided in the inpatient rehabilitation setting. This includes, but is not limited to , therapeutic activity, therapeutic exercise, neuromuscular re-education. This group is retrospectively collected, and will not include participants who had access to the BAT.
- Bimanual Arm Trainer: Participants who are prospectively enrolled, who are appropriate for BAT use. Participants will receive additional traditional occupational therapy interventions, as deemed appropriate by treating therapists.
  Interventions: Device: Bimanual Arm Trainer

INTERVENTIONS:
Device: Bimanual Arm Trainer — tabletop/desktop device that couples bilateral simultaneous upper extremity movement with virtual reality games or activities via computer monitor
  Groups: Bimanual Arm Trainer

SUMMARY:
Recent studies have shown that completing bilateral simultaneous movements during upper extremity practice may result in facilitation of coactivation and interhemispheric activation of both the ipsilesional and contralesional brain areas, with one limb entraining the other and enabling the limbs to function as a unit. Other research has proposed that the use of virtual-reality (VR) activities during treatment sessions can improve upper extremity function following stroke as it is motivating, challenging, offers external feedback that may facilitate motor learning, and allows for the "high-intensity, repetitious practice necessary to drive recovery". Coupling bilateral simultaneous upper extremity movement and virtual-reality activities is the Bimanual Arm Trainer (BAT), a non-powered mechanical device by which the non-paretic upper extremity moves the paretic arm. The purpose of this study is to determine the effectiveness of the Bimanual Arm Trainer (BAT) compared to traditional occupational therapy treatment sessions as these relate to upper extremity functional return following stroke, as measured by scores on the Action Research Arm Test (ARAT) and Upper Extremity Fugl-Meyer Assessment (UE-FMA) measures. The investigators plan to use retrospective data for a pre-implementation group, comparing this data to prospectively collected post-implementation data. ARAT scores are routinely collected and will be used for comparison between groups. UE-FMA measures are commonly used in this area of research, and will be taken to provide additional context for the post-implementation group.

DETAILED DESCRIPTION:
The medical charts of patients with a diagnosis of stroke will be reviewed retroactively to determine if there is a significant difference in improvement of upper extremity function (measured by ARAT and UE-FMA scores) following traditional occupational therapy services vs. use of the bimanual arm trainer. Medical charts of patients from November 2019 to November 2020 will be reviewed to obtain ARAT scores of patients who received traditional occupational therapy services. The Bimanual Arm Trainer was obtained in April 23, 2020; however, due to the pandemic, it was not able to be utilized until November 13, 2020. Patients from Review Board-approval onward will be assessed for ARAT and FMA-UE scores while using the device.

Duration: A minimum of 10 minutes for 3 separate sessions with Occupational Therapy for BAT participation. 15-30 minutes with Occupational Therapy (OT) within 3 days of admission and discharge for ARAT administration. The investigators anticipate that without mixed retrospective/prospective collection sample (post intervention application), the investigators will be able to reach the investigators' target participant number in 12 months after approval.

This study will not use a placebo or non-treatment group. The investigators will compare data retrospectively to patients who received standard care prior to the BAT being accessible within the investigators' rehabilitation department. Once the BAT was obtained and training occurred on the unit among staff members, the device was considered standard of care treatment to qualifying stroke patients; therefore, there is not a placebo group in the prospective portion of this study. Appropriate patient's will receive treatment sessions on the BAT regardless of participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute stroke.
* Score of <17 on admission ARAT.
* Participation ≥ 3 BAT training sessions.

Exclusion Criteria:

* Impaired cognition impacting ability to participate in virtual reality system
* Pain resulting in poor tolerance of range of motion.
* Impaired sitting balance or poor tolerance of sitting in upright posture in chair without armrests.
* Spasticity in the affected upper extremity Modified Ashworth Scale (MAS) of 3 or greater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with acute or sub-acute stroke, with upper extremity paresis, admitted to an Acute Inpatient Rehab (IRF/AIR) unit.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Change in Action Research Arm Test score | Within 72 hours of admission and up to 72 hours of discharge for all participants
  a standardized tool that assesses UE functional limitations based off of 19 action-based items. Scores range from a minimum of 0 to a maximum of 57 points, with higher scores reflecting greater upper extremity functioning.

SECONDARY OUTCOMES:
Change in Upper Extremity Fugl-Meyer Assessment score | Within 72 hours of admission and Up to 72 hours of discharge for all participants in the BAT group
  The UE-FMA is a body-functional level assessment of upper arm movement and sensation. Scores range from a minimum of o to a maximum of 66 points, with higher scores reflecting greater control of movement.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Babunovic, DPT, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Specialty Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No